CLINICAL TRIAL: NCT07328022
Title: Efficacy and Safety Study of the Etoricoxib/Betamethasone Combination Compared With Etoricoxib for the Treatment of Patients Diagnosed With an Acute Episode of Bursitis, Tendinitis, or Synovitis of the Shoulder, Elbow, Knee, or Ankle
Brief Title: Efficacy and Safety of Etoricoxib/Betamethasone Combination in Acute Bursitis, Tendinitis and Synovitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIL-30953-III-24(1)
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Bursitis; Tendinitis; Synovitis
Keywords: Bursitis; Tendinitis; Synovitis; Etoricoxib; Betamethasone; Acute Episode
MeSH Terms: conditions — Bursitis; Tendinopathy; Synovitis | interventions — Etoricoxib; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoricoxib + Betamethasone (Experimental): Administered orally, 1 tablet a day for 14 days.
  Interventions: Drug: Fixed Dose Etoricoxib + Betamethasone
- Etoricoxib (Active Comparator): Administered orally, 1 tablet a day for 14 days.
  Interventions: Drug: Monotherapy Etoricoxib

INTERVENTIONS:
Drug: Fixed Dose Etoricoxib + Betamethasone — One tablet of 90 mg / 0.25 mg a day, for 14 days
  Arms: Etoricoxib + Betamethasone
Drug: Monotherapy Etoricoxib — One tablet aog 90 mg a day, for 14 days
  Arms: Etoricoxib

SUMMARY:
Phase III, multicenter, prospective, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of a fixed-dose combination of etoricoxib/betamethasone compared with etoricoxib alone in patients with an acute episode of bursitis, tendinitis, or synovitis affecting the shoulder, elbow, knee, or ankle.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, prospective, randomized, double-blind, parallel-group study to compare the efficacy and safety of a fixed-dose combination of etoricoxib/betamethasone versus etoricoxib alone in patients with an acute episode of bursitis, tendinitis, or synovitis of the shoulder, elbow, knee, or ankle. Eligible participants will be randomized to receive either etoricoxib/betamethasone 90 mg/0.25 mg once daily for 14 days (Group A) or etoricoxib 90 mg once daily for 14 days (Group B). The study includes three visits (Day 1 baseline, Day 7 ± 2, Day 14 ± 2) and two follow-up calls (Day 3 ± 2 and Day 10 ± 2); investigators will collect medical history, perform physical examinations focused on the affected region, and review laboratory and diagnostic assessments as applicable. Pain intensity in the affected joint will be assessed using a Visual Analog Scale (VAS) during active movement and at rest at each visit/call, and daily by patients in a trained Patient Diary completed in the afternoon at the same time each day. Outcomes include changes from baseline in maximum pain (movement and rest) over 14 days, clinical improvement at Days 7 and 14 using the Clinical Global Impression scale, patient and investigator global assessments, and safety based on adverse events summarized by treatment group; rescue medication use (paracetamol 500 mg) and treatment adherence will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to participate in the study and provide written informed consent.
* Male or female.
* Age ≥ 18 years at study entry.
* Women of childbearing potential who use an acceptable contraceptive method (barrier, oral hormonal, injectable, subdermal), or women who are naturally postmenopausal or surgically sterile.
* Clinical diagnosis of an acute episode of tendinitis, bursitis, or synovitis of the shoulder, elbow, knee, or ankle, with onset within 7 days prior to the first dose of study medication.
* A score ≥ 40 mm on a 100-mm Visual Analog Scale (VAS) for maximum pain intensity during active movement, as reported by the patient at the time of study inclusion.
* In the opinion of the Principal Investigator or treating physician, the participant is an appropriate candidate for treatment with the investigational product.

Exclusion Criteria:

* Participation in another clinical study involving an investigational treatment, or participation in such a study within 4 weeks prior to study start.
* Patients whose participation could be influenced (e.g., employment relationship with the study site or sponsor, vulnerable populations, etc.).
* In the investigator's medical judgment, any disease that affects prognosis and prevents outpatient management, including but not limited to: terminal cancer, renal, cardiac, respiratory, or hepatic failure, mental illness, or scheduled surgical procedures or hospitalizations.
* History or presence of any disease or condition that, in the investigator's opinion, could pose a risk to the patient or confound the efficacy and safety evaluation of the investigational product, such as significant degenerative disease or an infectious process in the joints of interest.
* Fever: axillary temperature > 37.5°C within 2 days prior to or at the time of study inclusion.-
* Pregnant or breastfeeding patients.
* Contraindication to the study medications.
* History of allergic reaction to NSAIDs (non-steroidal anti-inflammatory drugs), paracetamol (acetaminophen), or known hypersensitivity to the study medications.
* Significant history of gastrointestinal disorders (e.g., gastric ulcer, Crohn's disease, ulcerative colitis, gastrointestinal bleeding, etc.).
* History of congestive heart failure (NYHA Class II-IV), established ischemic heart disease, peripheral arterial disease and/or cerebrovascular disease (including patients who have recently undergone coronary revascularization procedures or angioplasty).
* Treatment with corticosteroids within 1 month prior to study start.
* Treatment with NSAIDs within 48 hours prior to study start, except for cardioprotective-dose aspirin.
* Tendinitis or bursitis secondary to a systemic inflammatory disease, or synovitis secondary to hemophilia.
* History of harmful alcohol and/or drug use causing adverse health and social effects.
* Clinical suspicion of joint infection or another joint disease other than tendinitis, bursitis, or synovitis.
* History of chronic hepatic impairment (Child-Pugh A, B, and/or C).
* History of acute renal failure or chronic kidney disease (glomerular filtration rate < 30 mL/min/1.73 m²).
* Significant history of known coagulation disorders (e.g., von Willebrand disease, hemophilia, vitamin K deficiency, etc.) or use of anticoagulants.
* Oncology patients (except basal cell skin cancer or patients with cancer in remission) or patients with severe diseases that, in the investigator's opinion, have a poor prognosis or a life expectancy of less than 1 year, as well as mental illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Change in pain during active movement of the affected joint (VAS 100 mm) at Days 3, 7, 10, and 14 vs baseline, by treatment group. | Baseline and Days 3, 7, 10, and 14
  Pain intensity during active movement will be assessed using a 100-mm Visual Analog Scale (VAS) to determine whether the fixed-dose combination etoricoxib/betamethasone produces a greater reduction in pain compared with etoricoxib alone. Assessments will be obtained at baseline and at follow-up timepoints.
Number of participants with adverse events, and comparison of adverse event frequency and intensity, by treatment group. | Up to 14 days
  Safety will be assessed by comparing adverse events occurring during the study between treatment groups. Adverse events will be summarized using frequencies and percentages and classified according to seriousness/gravity, severity, and causality.

SECONDARY OUTCOMES:
Baseline sociodemographic, anthropometric, biochemical, and clinical characteristics, by treatment group. | Baseline
  Descriptive summary of participant characteristics at baseline by randomized group.
Daily change in maximum pain during active movement of the affected joint (VAS 100 mm) over 14 days vs baseline, by treatment group. | Daily through Day 14
  Patients will record daily VAS scores to estimate the magnitude of change from baseline in maximum pain during active movement throughout treatment.
Daily change in maximum pain at rest of the affected joint (VAS 100 mm) over 14 days vs baseline, by treatment group. | Daily through Day 14
  Patients will record daily VAS scores at rest to estimate the magnitude of change from baseline throughout treatment
Clinical improvement using the Clinical Global Impression (CGI) scale at Days 7 and 14 vs baseline, by treatment group. | Baseline, Day 7, and Day 14
  Clinical improvement will be evaluated using CGI (severity/improvement categories) at follow-up and compared with baseline by treatment group.
Change in Patient Global Assessment of current condition at Days 7 and 14 vs baseline, by treatment group. | Baseline, Day 7, and Day 14
  The Patient Global Assessment will be recorded and changes from baseline will be described by treatment group.
Proportion of patients by category on the Patient Global Assessment at Days 7 and 14 vs baseline, by treatment group. | Baseline, Day 7, and Day 14
  Changes in the proportion of patients reporting feeling very well, well, fair, poor, or very poor will be summarized by group.
Change in Investigator Global Assessment at Days 7 and 14 vs baseline, by treatment group. | Baseline, Day 7, and Day 14
  The Investigator Global Assessment will be recorded and changes from baseline will be described by treatment group.
Proportion of patients by category on the Investigator Global Assessment at Days 7 and 14 vs baseline, by treatment group. | Baseline, Day 7, and Day 14
  Changes in the proportion of participants classified as very well, well, fair, poor, or very poor by the investigator will be summarized by group.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Cordova Martinez, MD, Principal Investigator — Unidad de Medicina Especializada SMA SC; Pedro Abraham Garza Alvarez, MD, Principal Investigator — IECSI Clinical Research; Juan Luis Torres Mendez, MD, Principal Investigator — Clinical Research Institute S.C.; Yazmin Adriana Guerra Lopez, MD, Principal Investigator — Centro de Investigación Clínica de México S. de R.L. de C.V
Locations (1):
- Laboratorios Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov;5(11):1086-90. doi: 10.1111/j.1553-2712.1998.tb02667.x. PMID 9835471
- [Background] Bertin P, Behier JM, Noel E, Leroux JL. Celecoxib is as efficacious as naproxen in the management of acute shoulder pain. J Int Med Res. 2003 Mar-Apr;31(2):102-12. doi: 10.1177/147323000303100206. PMID 12760313
- [Background] Pincus T, Swearingen CJ, Luta G, Sokka T. Efficacy of prednisone 1-4 mg/day in patients with rheumatoid arthritis: a randomised, double-blind, placebo controlled withdrawal clinical trial. Ann Rheum Dis. 2009 Nov;68(11):1715-20. doi: 10.1136/ard.2008.095539. Epub 2008 Dec 15. PMID 19074913
- [Background] Pallay RM, Seger W, Adler JL, Ettlinger RE, Quaidoo EA, Lipetz R, O'Brien K, Mucciola L, Skalky CS, Petruschke RA, Bohidar NR, Geba GP. Etoricoxib reduced pain and disability and improved quality of life in patients with chronic low back pain: a 3 month, randomized, controlled trial. Scand J Rheumatol. 2004;33(4):257-66. doi: 10.1080/03009740410005728. PMID 15370723
- [Background] Matsumoto AK, Melian A, Mandel DR, McIlwain HH, Borenstein D, Zhao PL, Lines CR, Gertz BJ, Curtis S; Etoricoxib Rheumatoid Arthritis Study Group. A randomized, controlled, clinical trial of etoricoxib in the treatment of rheumatoid arthritis. J Rheumatol. 2002 Aug;29(8):1623-30. PMID 12180720
- [Background] Pisaniello HL, Fisher MC, Farquhar H, Vargas-Santos AB, Hill CL, Stamp LK, Gaffo AL. Efficacy and safety of gout flare prophylaxis and therapy use in people with chronic kidney disease: a Gout, Hyperuricemia and Crystal-Associated Disease Network (G-CAN)-initiated literature review. Arthritis Res Ther. 2021 Apr 28;23(1):130. doi: 10.1186/s13075-021-02416-y. PMID 33910619
- [Background] (EMA), E.M.A., Guideline on clinical development of fixed combination medicinal products. 2017.
- [Background] Rice JB, White AG, Scarpati LM, Wan G, Nelson WW. Long-term Systemic Corticosteroid Exposure: A Systematic Literature Review. Clin Ther. 2017 Nov;39(11):2216-2229. doi: 10.1016/j.clinthera.2017.09.011. Epub 2017 Oct 19. PMID 29055500
- [Background] la Torre LF, Franco-Gonzalez DL, Brennan-Bourdon LM, Molina-Frechero N, Alonso-Castro AJ, Isiordia-Espinoza MA. Analgesic Efficacy of Etoricoxib following Third Molar Surgery: A Meta-analysis. Behav Neurol. 2021 Sep 8;2021:9536054. doi: 10.1155/2021/9536054. eCollection 2021. PMID 34539935
- [Background] Watson DJ, Bolognese JA, Yu C, Krupa D, Curtis S. Use of gastroprotective agents and discontinuations due to dyspepsia with the selective cyclooxygenase-2 inhibitor etoricoxib compared with non-selective NSAIDs. Curr Med Res Opin. 2004 Dec;20(12):1899-908. doi: 10.1185/030079904X12681. PMID 15701208
- [Background] Petri M, Hufman SL, Waser G, Cui H, Snabes MC, Verburg KM. Celecoxib effectively treats patients with acute shoulder tendinitis/bursitis. J Rheumatol. 2004 Aug;31(8):1614-20. PMID 15290743
- [Background] Maquirriain J, Kokalj A. Management of acute Achilles tendinopathy: effect of etoricoxib on pain control and leg stiffness. Georgian Med News. 2013 Sep;(222):36-43. PMID 24099813
- [Background] Becker DE. Basic and clinical pharmacology of glucocorticosteroids. Anesth Prog. 2013 Spring;60(1):25-31; quiz 32. doi: 10.2344/0003-3006-60.1.25. PMID 23506281
- [Background] Han, S., Clinical pharmacology review for primary health care providers: II. Steroids. Transl Clin Pharmacol., 2015.
- [Background] Gómez Valdés, A., Y. Mendoza Cabrera, and L. Escalante Cambeaux, Sinovitis de rodilla, su tratamiento en el área terapéutica de la Facultad de Cultura Física "Nancy Uranga Romagoza". Podium. Revista de Ciencia y Tecnología en la Cultura Física, 2018. 13: p. 274-286.
- [Background] Tak PP, Breedveld FC. Current perspectives on synovitis. Arthritis Res. 1999;1(1):11-6. doi: 10.1186/ar4. Epub 1999 Oct 26. No abstract available. PMID 11094407
- [Background] Miranda H, Viikari-Juntura E, Martikainen R, Riihimaki H. A prospective study on knee pain and its risk factors. Osteoarthritis Cartilage. 2002 Aug;10(8):623-30. doi: 10.1053/joca.2002.0796. PMID 12479384
- [Background] van der Windt DA, Koes BW, Boeke AJ, Deville W, De Jong BA, Bouter LM. Shoulder disorders in general practice: prognostic indicators of outcome. Br J Gen Pract. 1996 Sep;46(410):519-23. PMID 8917870
- [Background] Green S, Buchbinder R, Hetrick S. Physiotherapy interventions for shoulder pain. Cochrane Database Syst Rev. 2003;2003(2):CD004258. doi: 10.1002/14651858.CD004258. PMID 12804509